CLINICAL TRIAL: NCT05483738
Title: The Impact of Mitochondrial Dysfunction on Human Bone Cell Metabolism and Remodelling
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Odense University Hospital (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Anja Lisbeth Frederiksen, MD, Ph.D, Clinical Professor, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S-20180170
Record Dates: First submitted 2022-07-22; First posted 2022-08-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Mitochondrial Diseases; Bone Remodeling Disorder
Keywords: m3243A>G; POLG; TWNK; Mitochondria
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Matched case-control study
Masking Description: Participants are masked with anonymized identifier (ID)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cases and controls (Other): Clinical assessment, blood samples, dual energy x-ray absorptiometry (DXA) scan, and assessment of bone marrow, and tetracycline labelled bone biopsy
  Interventions: Diagnostic Test: Clinical assessment, blood samples, bone marrow and bone biopsy

INTERVENTIONS:
Diagnostic Test: Clinical assessment, blood samples, bone marrow and bone biopsy — Assessment of blood samples, bone marrow and bone biopsy

SUMMARY:
Cell and mice studies suggest mitochondrial dysfunction may cause altered bone structure.

Hypothesis: Decreased mitochondrial energy production affects bone cell development and activity negatively.

Comparing humans with the mitochondrial DNA variant, m.3243A>G, pathogenic variants in POLG or TWNK genes to healthy controls, the aim is to evaluate the effect of mitochondrial dysfunction on: 1: bone-cell development and -activity in bone marrow stem cells and blood.

2: bone cell metabolism including glucose consumption. 3: bone structure assessed by electron microscopy and μCT scans of bone biopsies.

DETAILED DESCRIPTION:
Intact mitochondrial activity including adequate energy supplies is vital for metabolic active tissues i.e. skeletal muscle, heart and brain. The human skeleton represent an additional highly metabolically active tissue; nevertheless the significance of the mitochondrial role in human skeletal bone health may be further investigated.

Bone remodelling constitutes the coupled and continuous regenerative process of bone degradation by bone resorbing cells osteoclasts (OC) followed by formation of bone matrix by bone forming osteoblasts (OB). Quantitative imbalance between resorption and formation results in skeletal disorders with low bone mass including osteoporosis, and its increased risk of fragility fractures.

Mitochondria generate cellular energy adenosine triphosphate (ATP) through oxidative phosphorylation process (OXPHOS) in the respiratory chain (RC) with a secondary production of the deleterious by-products free radicals i.e. reactive oxygen species (ROS). Notably, mitochondria hold their own DNA (m.DNA), and RC subunits are encoded by m.DNA and nuclear DNA (n.DNA) genes, respectively. With ageing, deleterious somatic m.DNA mutations accumulate in skeletal muscle and heart, and somatic m.DNA mutations as well as inherited m.DNA or n.DNA mutations may result in mitochondrial dysfunction with impaired ATP production and accumulation of ROS. m.DNA mutations may impair brain, skeletal-, and cardiac muscle function, but the effects on human bone cell metabolism and remodelling are unknown. A recent study of a cohort of young individuals indicates that mitochondrial diseases pose a risk for bone fragility fractures.

Preclinical studies suggest that ATP and ROS regulate bone metabolism. The m.DNA number and mitochondrial activity increase to support differentiation from human skeletal (mesenchymal) stem cells (hMSC) to mature bone forming OBs. Inhibition of mitochondrial activity or increase in ROS levels suppress OB differentiation. Similarly, OCs are rich in mitochondria. Human OC cultures demonstrate that energy supplies for OC differentiation from their progenitors is based on OXPHOS while OC resorption activity relies on glycolysis.

In addition, emerging evidence suggest that metabolic plasticity i.e. regulation of glycolysis, OXPHOS, and pyruvate levels, contribute to regulation of OB and OC differentiation.

Receptor activator of nuclear factor kappa-Beta ligand (RANKL) secreted by OBs activates OC resorption. In mice, RANKL stimulation of bone marrow OC progenitors increases intracellular levels of ROS, which stimulates OC differentiation and bone resorption in-vitro. Further, ROS inhibits the wingless-type (Wnt) signalling pathway with attenuation of osteoblastogenesis and decreased bone formation.

Furthermore, mice with mutations in the n.DNA encoded proof reading domain of m.DNA polymerase POLG (PolgA-/-) accumulate m.DNA mutations, and present with premature ageing phenotype including low bone mass. In addition, deficiency of the n.DNA encoded mitochondrial transcription factor (TFAM) causes ATP depletion, and mice with TFAM deficient OCs have increased OC activity and augmented bone resorption. Opposite, global loss of NADH (nicotinamide-adenine dinucleotide) ubiquinone oxidoreductase Fe-S protein 4 (NDUFS4) a subunit in RC complex 1 impairs bone resorption, and (ndufs4-/-) mice present with increased bone mineral density (BMD) and an apparent osteopetrosis bone phenotype.

The aim is to study bone cell phenotype in patients with rare mitochondrial disease Carriers of MT-TL1 m.3243A>G (MIM: 590050).The gene encodes the transcription factor tRNALeu(UUA/UUG) and m.3243A>G weakens the assembly of RC complex with a secondary impaired ATP production. The phenotype is, in part associated with the m.3243A>G mutation burden i.e. level of heteroplasmy (percentage of m.3243A>G/wildtype m.DNA). The study group also includes carriers of mutations in the nuclear encoded POLG (MIM: 174763) and TWNK (MIM: 606075).

Hypothesis: Impaired mitochondrial function affects human bone cell -differentiation, -metabolism, and -activity leading to impaired bone formation and bone fragility.

Aim: To determine if carriers of inherited mitochondrial mutations i.e. mitochondrial dysfunction, ATP depletion and secondary increase in ROS lead to change in:

1. In-vitro OB differentiation-rate, OB activity and bone formation.
2. In-vitro OC differentiation-, OC activity and higher overall bone resorption.
3. In-vivo changes in tissues level dynamics of bone formation and - resorption as examined in iliac crest bone biopsies.

Design, Participants and Methods: Cross-sectional case-control study including subjects (>18 years) carrying one of the following mutations:

1. MT-TL1 m.3243A>G
2. POLG mutation
3. TWNK

N=10 cases with each pathogenic genetic variant and equal number of controls (n=30) matched on sex, age and BMI.

ELIGIBILITY:
Inclusion Criteria - cases:

* Genetic diagnosis with: MT-TL1 m.3243A>G, or POLG variant, het or TWNK variant, het, > 18 years
* Signed informed consent

Inclusion Criteria - controls:

* Healthy subjects matched on age and gender > 18 years
* Signed informed consent

Exclusion Criteria:

* Renal (creatinine > 90 µmol/l)
* Liver dysfunction (AST > 3 times the upper limit)
* Medical treatment influencing bone metabolism (oral corticosteroid <12 weeks, anti-osteoporosis treatment, sex steroids, anti-convulsants)
* Pregnancy
* Excessive consumption of alcohol
* Treatment with anticoagulants
* Pre-existing coagulopathy
* Allergy to lidocaine, morphine or diazepam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Extracellular acidification rate (ECAR) (mpH/min) | Up to 12 weeks
  Measurement of ECAR in human bone marrow skeletal (mesenchymal) stem cells (hBM-MSCs), osteoblasts (OB) and osteoclasts (OC)
Oxygen consumption rate (OCR) (mpMol/min) | Up to 12 weeks
  Measurement of OCR in hBM-MSCs, OBs and OCs
Growth rate (number of cells) | Up to 12 weeks
  Growth rate of of OBs and OCs

SECONDARY OUTCOMES:
Bone growth rate (µm/day) | Up to 4 weeks
  Histomophometric measurements of bone growth in tetracycline labeled bone biopsy
Histomorphometric | Up to 4 weeks
  Histomophometric studies of bone biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Anja L Frederiksen, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Dept. of Clinical Genetics, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorman GS, Chinnery PF, DiMauro S, Hirano M, Koga Y, McFarland R, Suomalainen A, Thorburn DR, Zeviani M, Turnbull DM. Mitochondrial diseases. Nat Rev Dis Primers. 2016 Oct 20;2:16080. doi: 10.1038/nrdp.2016.80. PMID 27775730
- [Background] Seeman E, Delmas PD. Bone quality--the material and structural basis of bone strength and fragility. N Engl J Med. 2006 May 25;354(21):2250-61. doi: 10.1056/NEJMra053077. No abstract available. PMID 16723616
- [Background] Bartell SM, Kim HN, Ambrogini E, Han L, Iyer S, Serra Ucer S, Rabinovitch P, Jilka RL, Weinstein RS, Zhao H, O'Brien CA, Manolagas SC, Almeida M. FoxO proteins restrain osteoclastogenesis and bone resorption by attenuating H2O2 accumulation. Nat Commun. 2014 Apr 30;5:3773. doi: 10.1038/ncomms4773. PMID 24781012
- [Background] Andreasen CM, Ding M, Overgaard S, Bollen P, Andersen TL. A reversal phase arrest uncoupling the bone formation and resorption contributes to the bone loss in glucocorticoid treated ovariectomised aged sheep. Bone. 2015 Jun;75:32-9. doi: 10.1016/j.bone.2015.02.014. Epub 2015 Feb 14. PMID 25689083
- [Background] Kim SJ, Mehta HH, Wan J, Kuehnemann C, Chen J, Hu JF, Hoffman AR, Cohen P. Mitochondrial peptides modulate mitochondrial function during cellular senescence. Aging (Albany NY). 2018 Jun 10;10(6):1239-1256. doi: 10.18632/aging.101463. PMID 29886458
- [Background] Sinha K, Das J, Pal PB, Sil PC. Oxidative stress: the mitochondria-dependent and mitochondria-independent pathways of apoptosis. Arch Toxicol. 2013 Jul;87(7):1157-80. doi: 10.1007/s00204-013-1034-4. Epub 2013 Mar 30. PMID 23543009
- [Background] Meissner C, Bruse P, Mohamed SA, Schulz A, Warnk H, Storm T, Oehmichen M. The 4977 bp deletion of mitochondrial DNA in human skeletal muscle, heart and different areas of the brain: a useful biomarker or more? Exp Gerontol. 2008 Jul;43(7):645-652. doi: 10.1016/j.exger.2008.03.004. Epub 2008 Mar 20. PMID 18439778
- [Background] Lee HC, Wei YH. Oxidative stress, mitochondrial DNA mutation, and apoptosis in aging. Exp Biol Med (Maywood). 2007 May;232(5):592-606. PMID 17463155
- [Background] Hayashi G, Cortopassi G. Oxidative stress in inherited mitochondrial diseases. Free Radic Biol Med. 2015 Nov;88(Pt A):10-7. doi: 10.1016/j.freeradbiomed.2015.05.039. Epub 2015 Jun 12. PMID 26073122
- [Background] Gandhi SS, Muraresku C, McCormick EM, Falk MJ, McCormack SE. Risk factors for poor bone health in primary mitochondrial disease. J Inherit Metab Dis. 2017 Sep;40(5):673-683. doi: 10.1007/s10545-017-0046-2. Epub 2017 Apr 27. PMID 28451918
- [Background] Chen CT, Shih YR, Kuo TK, Lee OK, Wei YH. Coordinated changes of mitochondrial biogenesis and antioxidant enzymes during osteogenic differentiation of human mesenchymal stem cells. Stem Cells. 2008 Apr;26(4):960-8. doi: 10.1634/stemcells.2007-0509. Epub 2008 Jan 24. PMID 18218821
- [Background] Gao J, Feng Z, Wang X, Zeng M, Liu J, Han S, Xu J, Chen L, Cao K, Long J, Li Z, Shen W, Liu J. SIRT3/SOD2 maintains osteoblast differentiation and bone formation by regulating mitochondrial stress. Cell Death Differ. 2018 Feb;25(2):229-240. doi: 10.1038/cdd.2017.144. Epub 2017 Sep 15. PMID 28914882
- [Background] Brown D, Breton S. Mitochondria-rich, proton-secreting epithelial cells. J Exp Biol. 1996 Nov;199(Pt 11):2345-58. doi: 10.1242/jeb.199.11.2345. PMID 9114500
- [Background] Lemma S, Sboarina M, Porporato PE, Zini N, Sonveaux P, Di Pompo G, Baldini N, Avnet S. Energy metabolism in osteoclast formation and activity. Int J Biochem Cell Biol. 2016 Oct;79:168-180. doi: 10.1016/j.biocel.2016.08.034. Epub 2016 Aug 30. PMID 27590854
- [Background] Arnett TR, Orriss IR. Metabolic properties of the osteoclast. Bone. 2018 Oct;115:25-30. doi: 10.1016/j.bone.2017.12.021. Epub 2017 Dec 21. PMID 29274806
- [Background] Lee NK, Choi YG, Baik JY, Han SY, Jeong DW, Bae YS, Kim N, Lee SY. A crucial role for reactive oxygen species in RANKL-induced osteoclast differentiation. Blood. 2005 Aug 1;106(3):852-9. doi: 10.1182/blood-2004-09-3662. Epub 2005 Apr 7. PMID 15817678
- [Background] Garrett IR, Boyce BF, Oreffo RO, Bonewald L, Poser J, Mundy GR. Oxygen-derived free radicals stimulate osteoclastic bone resorption in rodent bone in vitro and in vivo. J Clin Invest. 1990 Mar;85(3):632-9. doi: 10.1172/JCI114485. PMID 2312718
- [Background] Almeida M, Han L, Martin-Millan M, O'Brien CA, Manolagas SC. Oxidative stress antagonizes Wnt signaling in osteoblast precursors by diverting beta-catenin from T cell factor- to forkhead box O-mediated transcription. J Biol Chem. 2007 Sep 14;282(37):27298-27305. doi: 10.1074/jbc.M702811200. Epub 2007 Jul 10. PMID 17623658
- [Background] Trifunovic A, Wredenberg A, Falkenberg M, Spelbrink JN, Rovio AT, Bruder CE, Bohlooly-Y M, Gidlof S, Oldfors A, Wibom R, Tornell J, Jacobs HT, Larsson NG. Premature ageing in mice expressing defective mitochondrial DNA polymerase. Nature. 2004 May 27;429(6990):417-23. doi: 10.1038/nature02517. PMID 15164064
- [Background] Miyazaki T, Iwasawa M, Nakashima T, Mori S, Shigemoto K, Nakamura H, Katagiri H, Takayanagi H, Tanaka S. Intracellular and extracellular ATP coordinately regulate the inverse correlation between osteoclast survival and bone resorption. J Biol Chem. 2012 Nov 2;287(45):37808-23. doi: 10.1074/jbc.M112.385369. Epub 2012 Sep 17. PMID 22988253
- [Background] Jin Z, Wei W, Yang M, Du Y, Wan Y. Mitochondrial complex I activity suppresses inflammation and enhances bone resorption by shifting macrophage-osteoclast polarization. Cell Metab. 2014 Sep 2;20(3):483-98. doi: 10.1016/j.cmet.2014.07.011. Epub 2014 Aug 14. PMID 25130399
- [Background] Varanasi SS, Francis RM, Berger CE, Papiha SS, Datta HK. Mitochondrial DNA deletion associated oxidative stress and severe male osteoporosis. Osteoporos Int. 1999;10(2):143-9. doi: 10.1007/s001980050209. PMID 10501795
- [Background] Kato H, Han X, Yamaza H, Masuda K, Hirofuji Y, Sato H, Pham TTM, Taguchi T, Nonaka K. Direct effects of mitochondrial dysfunction on poor bone health in Leigh syndrome. Biochem Biophys Res Commun. 2017 Nov 4;493(1):207-212. doi: 10.1016/j.bbrc.2017.09.045. Epub 2017 Sep 9. PMID 28899781
- [Background] Langdahl JH, Frederiksen AL, Hansen SJ, Andersen PH, Yderstraede KB, Duno M, Vissing J, Frost M. Mitochondrial Point Mutation m.3243A>G Associates With Lower Bone Mineral Density, Thinner Cortices, and Reduced Bone Strength: A Case-Control Study. J Bone Miner Res. 2017 Oct;32(10):2041-2048. doi: 10.1002/jbmr.3193. Epub 2017 Jul 18. PMID 28603900
- [Background] van den Ouweland JM, Lemkes HH, Ruitenbeek W, Sandkuijl LA, de Vijlder MF, Struyvenberg PA, van de Kamp JJ, Maassen JA. Mutation in mitochondrial tRNA(Leu)(UUR) gene in a large pedigree with maternally transmitted type II diabetes mellitus and deafness. Nat Genet. 1992 Aug;1(5):368-71. doi: 10.1038/ng0892-368. PMID 1284550
- [Background] Sasarman F, Antonicka H, Shoubridge EA. The A3243G tRNALeu(UUR) MELAS mutation causes amino acid misincorporation and a combined respiratory chain assembly defect partially suppressed by overexpression of EFTu and EFG2. Hum Mol Genet. 2008 Dec 1;17(23):3697-707. doi: 10.1093/hmg/ddn265. Epub 2008 Aug 27. PMID 18753147
- [Background] Frederiksen AL, Andersen PH, Kyvik KO, Jeppesen TD, Vissing J, Schwartz M. Tissue specific distribution of the 3243A->G mtDNA mutation. J Med Genet. 2006 Aug;43(8):671-7. doi: 10.1136/jmg.2005.039339. Epub 2006 Feb 20. PMID 16490799
- [Background] Langdahl JH, Larsen M, Frost M, Andersen PH, Yderstraede KB, Vissing J, Duno M, Thomassen M, Frederiksen AL. Lecocytes mutation load declines with age in carriers of the m.3243A>G mutation: A 10-year Prospective Cohort. Clin Genet. 2018 Apr;93(4):925-928. doi: 10.1111/cge.13201. PMID 29266179
- [Background] Jafari A, Qanie D, Andersen TL, Zhang Y, Chen L, Postert B, Parsons S, Ditzel N, Khosla S, Johansen HT, Kjaersgaard-Andersen P, Delaisse JM, Abdallah BM, Hesselson D, Solberg R, Kassem M. Legumain Regulates Differentiation Fate of Human Bone Marrow Stromal Cells and Is Altered in Postmenopausal Osteoporosis. Stem Cell Reports. 2017 Feb 14;8(2):373-386. doi: 10.1016/j.stemcr.2017.01.003. Epub 2017 Feb 2. PMID 28162997
- [Background] Abdallah BM, Ditzel N, Kassem M. Assessment of bone formation capacity using in vivo transplantation assays: procedure and tissue analysis. Methods Mol Biol. 2008;455:89-100. doi: 10.1007/978-1-59745-104-8_6. PMID 18463812
- [Background] Soe K, Delaisse JM. Glucocorticoids maintain human osteoclasts in the active mode of their resorption cycle. J Bone Miner Res. 2010 Oct;25(10):2184-92. doi: 10.1002/jbmr.113. PMID 20499345